CLINICAL TRIAL: NCT07137273
Title: Optimizing Dimensions of Reinforcement to Enhance Behavioral Interventions
Brief Title: Optimizing Dimensions of Reinforcement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Collaborators: Oakland University (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, John Michael Falligant, Assistant Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R21HD113881 (NIH)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Intellectual Disabilities (F70-F79); Autism
Keywords: Operant Conditioning; Neurodevelopmental disorders; Behavioral interventions
MeSH Terms: conditions — Intellectual Disability; Autistic Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: All participants receive the same sequence of experimental conditions. The design allows for within-subject comparisons across phases of the intervention to evaluate changes in operant responding under different schedule arrangements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm: Manipulation of Reinforcement Schedules (Experimental): Participants will complete an operant conditioning task in which reinforcement schedules are systematically manipulated to evaluate changes in response patterns. All participants receive the same sequence of experimental conditions, which involve varying the availability and distribution of points exchangeable for preferred items or activities. No health-related treatment is provided; the procedures are designed to examine basic behavioral processes related to reinforcement dynamics.
  Interventions: Behavioral: Operant Conditioning Tasks with Reinforcement Manipulations

INTERVENTIONS:
Behavioral: Operant Conditioning Tasks with Reinforcement Manipulations — This behavioral intervention involves structured operant conditioning tasks. Reinforcement parameters (e.g., schedule arrangement, magnitude, and probability) are systematically manipulated to evaluate their effects on behavioral allocation. The primary objective is to assess how variations in reinforcement contingencies influence choice patterns. The procedures are designed to examine fundamental behavioral processes rather than to provide therapeutic benefit.

SUMMARY:
This study is designed to better understand how certain features of reinforcement affect learning and motivation in individuals with intellectual and developmental disabilities (IDD). Participants will take part in a series of structured teaching sessions that involve simple tasks and reward-based feedback. By changing the timing and amount of rewards, we aim to learn how these factors influence the ability to acquire and maintain new skills. This information may help improve behavioral interventions for individuals with IDD in the future. The study does not involve medications or procedures intended to change participants' health status.

DETAILED DESCRIPTION:
This study examines how key parameters of reinforcement-specifically the timing and amount of rewards-affect learning, motivation, and performance in individuals with intellectual and developmental disabilities (IDD). The experimental design is informed by the Mathematical Principles of Reinforcement (MPR), a quantitative framework for understanding the relationship between reinforcement schedules and behavior.

Participants will complete tabletop tasks in a controlled setting. Tasks are designed to be simple and accessible, such as pressing a button or selecting a picture, and correct responses will earn small rewards. Across sessions, we will systematically vary reinforcement parameters, including inter-reinforcement interval and reinforcer magnitude, to evaluate their effects on response rate, accuracy, and persistence.

This is a Basic Experimental Studies with Humans (BESH) clinical trial, meaning the interventions are intended to understand fundamental behavioral processes, not to produce direct clinical benefit. The data will be analyzed using statistical models derived from MPR to identify which reinforcement dimensions are most effective in maintaining high rates of responding. The results may help refine behavior intervention strategies for individuals with IDD by providing an evidence-based understanding of how to optimize reinforcement delivery.

ELIGIBILITY:
Inclusion Criteria:

At least 6 years of age

Documented neurodevelopmental condition

Engagement in problem behavior (e.g., aggression, self-injury, property destruction) that can be measured during study sessions

Ability to follow simple instructions

Ability to participate in tabletop choice-based tasks

Availability to complete all scheduled study sessions

Provision of informed consent by participant or legally authorized representative

Exclusion Criteria:

Severe sensory or motor impairments that would prevent participation in tabletop tasks

Current or recent participation (within the past 30 days) in another interventional behavioral research study that could interfere with study outcomes

Medical or behavioral conditions judged by investigators to pose a safety risk or interfere with data collection

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in rate of behavior across schedules | 3 months
  Number of target responses allocated emitted during experimental sessions in which reinforcement parameters (e.g., schedule arrangement, magnitude, and probability) are systematically varied. This measure will be derived from response data recorded during operant conditioning tasks. Changes in allocation patterns will be compared across schedule conditions to assess the effect of reinforcement manipulations.

CONTACTS AND LOCATIONS:
Overall Officials: John M Falligant, PhD, Principal Investigator — Auburn University
Locations (3):
- United States (3):
  - Center for Autism Research, Treatment, and Training, Auburn, Alabama
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Oakland University, Rochester Hills, Michigan

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and confidentiality, only aggregate data and summary results will be disseminated through publications, presentations, and ClinicalTrials.gov.

DOCUMENTS (1):
  • Informed Consent Form (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT07137273/ICF_000.pdf